

# TRIAL STATISTICAL ANALYSIS PLAN

C28709494-03

**BI Trial No.:** 1368-0010

**Title:** Proof-of-concept study of BI 655130 add-on treatment in patients

with mild-to-moderately active ulcerative colitis during TNF

inhibitor therapy

Including Protocol Amendment 3 [c11253289-04]

Investigational

**Product:** 

BI 655130

Responsible trial statisticians:

Phone: Fax:

**Date of statistical** 

04 March 2020 REVISED

analysis plan:

Version: 3.0

**** 

#### Proprietary confidential information

© 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

#### 1. **TABLE OF CONTENTS**

| TITLE PA | GE1 |
|--------------|------------------------------------------------|
| 1. | TABLE OF CONTENTS2 |
| LIST OF | ΓABLES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY10 |
| 5.<br>5.1 | ENDPOINTS12 PRIMARY ENDPOINT12 |
| 5.2<br>5.2.1 | SECONDARY ENDPOINTS 12 |
| 5.2.2 | Key secondary endpoints |
| 6. | GENERAL ANALYSIS DEFINITIONS18 |
| 6.1 | TREATMENTS |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS |
| 6.3 | SUBJECT SETS ANALYSED |
| 6.5 | POOLING OF CENTRES |
| 6.6<br>6.6.1 | HANDLING OF MISSING DATA AND OUTLIERS |
| 6.6.2 | Efficacy data 33 |
| 6.6.3 | Safety data 34 |
| 6.6.4 | PK data 34 |
| 6.6.5 | Biomarker data |
| 6.6.6 | Time since first diagnosis |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS35 |
| 7.<br>7.1 | PLANNED ANALYSIS |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION41 |
| 7.3 | TREATMENT COMPLIANCE 42 |

| 7.4.1 Primary analysis of the primary endpoint |
|---|
| primary endpoint 43 7.5 SECONDARY ENDPOINTS 45 7.5.1 Key secondary endpoints 45 |
| 7.5 SECONDARY ENDPOINTS |
| 7.5.1 Key secondary endpoints |
| 7.5.1 Key secondary endpoints |
| = ======= ; water ; or or are in a second for the point of infilling of infilling infillin |
| 7.5.1.2 Sensitivity analysis, subgroup analysis, exploratory analysis of the key |
| secondary endpoint(s) 45 |
| 7.5.2 (Other) Secondary endpoints |
| ( Other ) Secondary Chaptering Management ( ) |
| 7.7 EXTENT OF EXPOSURE 49 |
| 7.8 SAFETY ANALYSIS |
| 7.8.1 Adverse events |
| 7.8.2 Laboratory data |
| 7.8.3 Vital signs |
| 7.8.4 ECG |
| 7.8.5 Others |
| 8. REFERENCES |
| 10 HISTORY TARLE 67 |

# LIST OF TABLES

| Table 6.1: 1 | Flow chart of analysis phases | 18 |
|---|---|---|
| Table 6.2: 1 | Handling of iPDs | 20 |
| Table 6.3: 1 | Subject sets analysed | 30 |
| Table 6.7: 1 | Time windows for assignment of efficacy, safety lab, vital signs and | |
| | biomarker to visits for statistical analysis | 36 |
| Table 7.1: 1 | Categories for summary of continuous variables | 40 |
| Table 7.4.2: 1 | Summary of all analyses to be performed for the primary endpoint | 44 |
| Table 7.5.2: 1 | Summary of all analyses to be performed for the secondary endpoints | 46 |
| Table 7.8.1: 1 | Project MEDDRA search criteria for User Defined Adverse Events | |
| | Concepts | 52 |
| Table 10: 1 | History table | 67 |

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|--------|--------------------------------------------------|
| ADA | Anti-drug antibodies |
| ADS | Analysis dataset |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALQ | Above limit of quantification |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BM-SAP | Biomarker Statistical Analysis Plan |
| BMI | Body mass index |
| BRAVE | BI RAVE® |
| BRPM | Blinded Report Planning Meeting |
| CARE | Clinical data analysis and reporting environment |
| CHI3L1 | Faecal chitinase 3-like-1 |
| CR | Clinical remission |
| CRF | Case report form |
| CRP | C-reactive protein |
| CTC | Common Terminology Criteria |
| CTP | Clinical trial protocol |
| CTR | Clinical trial report |
| DBLM | Database lock meeting |
| DMC | Data Monitoring Committee |
| DNA | Deoxyribonucleic acid |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDC | Electronic Data Capture |
| EMA | European Medicines Agency |
| EOS | End of Study |
| EOT | End of treatment |

| Term | Definition / description |
|---|---|
| ES | Enrolled set |
| EudraCT | European union drug regulating authorities clinical trials |
| FAS | Full analysis set |
| FLF | Faecal lactoferrin |
| F-NGAL | Faecal neutrophil gelatinase-associated lipocalin |
| HMGB1 | High-mobility group box 1 protein |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| IL | Interleukin |
| iPD | Important protocol deviation |
| IRT | Interactive response technology |
| KM | Kaplan-Meier |
| LD | Day of Last dose/infusion received |
| LLOQ | Lower limit of quantification |
| LOQ | Limit of quantification |
| MCS | Mayo Clinical Score |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mESS | Modified Endoscopic Subscore |
| MPO | myeloperoxidase |
| MQRM | Medical quality review meeting |
| NOA | Not analysed |
| NOP | No peak detectable |
| NOR | No valid result |
| NOS | No sample available |
| NRI | Non response imputation |
| NRI-IR | Non Response Imputation including rescue medication |
| OC | Observed cases |
| OC-IR | Observed cases including values after rescue medication |
| OR | Original results |
| pCR | Partial MCS remission |
| PD | Pharmacodynamic(s) |
| PG | Pharmacogenomic(s) |

| Term | Definition / description |
|------|---------------------------------------|
| PGA | Physician Global Assessment |
| PK | Pharmacokinetic(s) |
| PPS | Per protocol set |
| PT | Preferred Term |
| PD | Protocol Deviation |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| RAGe | Report appendix generator |
| RBS | Rectal Bleeding Subscore |
| RCTC | Rheumatology Common Toxicity Criteria |
| REP | Residual effect period |
| RS | Randomized set |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDL | Subject data listing |
| SFS | Stool Frequency Score |
| SMQ | Standardised MedDRA query |
| SOC | System Organ Class |
| tCR | Total clinical remission |
| TCM | Trial Clinical Monitor |
| TSAP | Trial statistical analysis plan |
| ULN | Upper limit of normal range |
| ULOQ | Upper limit of quantification |
| VAS | Visual analogue scale |

**Trial No: 1368-0010 – 3.0 (Final)** 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

The screening of patients in the study was prematurely discontinued on February 4<sup>th</sup>, 2020. At that time, 22 patients had been randomized into the study and 15 patients had completed the trial. Five patients had completed through Week 12, but were still ongoing in the trial, and another two patients had not yet completed Week 12 and were still ongoing in the trial. There were no patients in the screening period. A decision was made that an early interim analysis of the Week 12 data would be done in order to discuss the results with both internal and external experts allowing for an early decision on the future of the project to be made.

The data cut-off for the interim snapshot of the database is February 4<sup>th</sup>, 2020. Of the five patients who have already completed Week 12 but are still ongoing, all five of them completed Week 12 prior to this cut-off date, leaving a total of 20 patients available for the interim analysis. The strategy for data cleaning in preparation for the interim snapshot of the database will be specified in a separate data cleaning plan.

The following data reporting strategy for safety and efficacy (along with any PK, ADA, and biomarker data which is available) is planned:

- A selection of data up to the Week 12 visit is to be summarized (including, at a minimum, the primary and secondary endpoints, as well as adverse event data). As a consequence of trial termination and of the need for a rapid decision on the future of the project, this analysis will be performed using the data of the 20 patients who have completed/discontinued through Week 12 prior to the cut-off date

For further details on the subject sets thus defined, refer to Section 6.3. For further details on the data to be included into the Week 12 analysis, refer to Table 6.7: 1. Further specification on the safety summaries to be performed at the time of the interim database snapshot are specified in Section 7.8.1. A logistics and access plan, which will describe any measures used to protect the blind and integrity of the ongoing trial will be finalized prior to database snapshot and treatment unblinding.

In accordance with the CTP, a second interim database snapshot will be performed once all randomized patients complete/discontinue through Week 12. At this time, all displays as

## **Boehringer Ingelheim**

**Trial No: 1368-0010 – 3.0 (Final)** 

**** 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

described in this TSAP will be produced. The results from this analysis will be used for potential authority interactions, if applicable.

A final analysis of the trial will be performed once all patients have completed the trial. For more details, please refer to Section 6.3.

Study data will be stored in a trial database within the BRAVE system.

The statistical analyses will be performed within the validated working environment CARE, including ), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses stated in the CTP (latest version) will be performed as planned with the following adaptations.

For within-project consistency, the following efficacy endpoints were modified, added or renamed.

The further endpoint "Clinical response" and "Time to flare" were modified as follows:

- Clinical response (total MCS decrease from baseline ≥3 points, and by ≥30%; AND RBS decrease from baseline by ≥1 point, or abs. ≤1) at Week 8 and at Week 12
- Time to flare was modified as time to suspected flare (increase in partial MCS by ≥2 from nadir)

The following endpoints were added to the list of further endpoints:

- Partial MCS response (Partial MCS (i.e. excluding mESS) decrease from baseline ≥2 points; AND RBS decrease from baseline by ≥1 point, or absolute value ≤1) over time
- Complete remission (Robarts Histology Index  $\leq 6$  and mESS=0) at Weeks 8 and 12
- Endoscopic remission (mESS=0) at Week 8 and at Week 12
- Percent change in faecal lactoferrin (FLF) at all measured time points as compared to baseline
- Change from baseline in SFS by visit (calculated as the average of the last 3 SFS measurements used in the derivation of the partial Mayo score)
- Change from baseline in RBS by visit (calculated as the average of the last 3 RBS measurements used in the derivation of the partial Mayo score)

The following endpoints have been renamed as below (see also Table 9.2.5: 1):

### Primary endpoint:

 "Mucosal healing" at Week 12 has been renamed "Endoscopic improvement" at Week 12

### **Secondary endpoints:**

- "Clinical remission" at Week 12 has been renamed "Total clinical remission (tCR)" at Week 12
- "Modified clinical remission" at Week 12 has been renamed "Clinical remission (CR)" at Week 12

## **Further endpoints:**

- "Clinical remission" at Week 8 has been renamed "Total clinical remission (tCR)" at Week 8
- "Modified clinical remission" at Week 8 has been renamed "Clinical remission (CR)" at Week 8

• "Partial clinical remission" at Week 8 and at Week 12 has been renamed "Partial MCS remission (pCR)" at Week 8 and at Week 12

Subsets of the subject sets (see Section 6.3) are now defined which include only those patients who completed/discontinued through Week 12 prior to the cut-off date February 4th, 2020. These subsets will be used for the reporting of the outputs at the time of the first interim database snapshot.

The Reeve method for calculating confidence intervals was removed from the analysis plan in <u>Section 7</u> due to low enrollment.

The subgroup analysis was expanded to include the concomitant use of steroids (yes/no) and prior TNFi failure (yes/no) (see Section 6.4).

### 5. ENDPOINTS

For all endpoints and unless explicitly specified otherwise, Week 8 refers to visit V5 using extended time windows as defined in Table 6.7: 1.

For all endpoints and unless explicitly specified otherwise, Week 12 refers to EOT visit using extended time windows as defined in Table 6.7: 1.

For handling of missing data and corresponding sensitivity analyses, see <u>Section 6.6</u>.

#### 5.1 PRIMARY ENDPOINT

Endoscopic improvement (MCS mESS  $\leq$ 1) at Week 12 is the primary endpoint.

Derivation of the mESS is described in Section 9.2: 1.

#### 5.2 SECONDARY ENDPOINTS

### 5.2.1 Key secondary endpoints

Not applicable – there are no key secondary endpoints for this trial.

### 5.2.2 **Secondary endpoints**

The secondary endpoints are listed below.

- Treatment emerging adverse events
- Total Clinical remission (tCR) based on Mayo score (total MCS ≤2 points, and all subscores ≤1 point) at Week 12
- Histological remission (Robarts (RHI) score ≤6) at Week 12
- Clinical remission (CR) based on Mayo score (total modified MCS ≤2 and: RBS =0, SFS =0 or 1 and drop ≥1 from baseline, AND mESS ≤1) at Week 12

Derivation of tCR, CR, and Histological remission is described in Section 9.2.













### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on the treatment to be administered, assignment to treatment, and selection of dose, see Section 4 of the CTP.

All patients will receive either intravenous doses of 1200mg of BI 655130 solution for infusion (at Weeks 0, 4 and 8), or placebo.

The following study phases are defined:

Table 6.1: 1 Flow chart of analysis phases

| Study analysis phase | Description | Start (included) | End (included) |
|---|---|---|---|
| Screening phase | Screening | Earliest of: i) Date of informed consent; ii) first screening procedure | Date/time of start of infusion of first study drug minus 1 minute. |
| Treatment phase & Residual effects | On-treatment period | Date/time of start of infusion of first study drug (Day 1) | Date of end of infusion of last<br>study drug + 140 days at 11:59 |
| period (REP) | 1 | | p.m. |
| Follow-up <sup>1</sup> phase | Off-treatment period | Date of end of infusion of last study drug + 141 days at 12:00 a.m. | Latest of: i) Date of EOS visit (Week 36 visit); ii) last contact date on End of Study page at 11:59 p.m. |

Dates are defined individually per patient. If more than one date is associated with a specific visit, measurements associated with a specific date are assigned to a study analysis phase according to the rules specified in the table. An analysis phase will not extend beyond the start date of the following phase.

The first interim database snapshot analysis will be performed based on the randomized patients who have completed/discontinued through the planned first 12 weeks of the trial up to the cut-off date, February 4th, 2020. For a description of the subject sets to be analysed, see Section 6.3. The following data will be used in this analysis:

• Selected summaries of the 12-week data will be performed up to the minimum of the (analysis-specific data cut-off; study day 99), unless otherwise specified.

The second interim database snapshot, to be performed once all randomized patients have completed/discontinued through the planned first 12 weeks of the trial (per CTP specification), will use the following data:

• All 12 weeks of data will be summarized up to the minimum of the (analysis-specific data cut-off; study day 99), unless otherwise specified.

The final analysis of the trial will be performed once all patients have completed the planned 36 weeks of trial; results will be summarized including all on-treatment data from the trial.

<sup>&</sup>lt;sup>1</sup> The off-treatment period (i.e. Follow-up phase) only exists if the trial completion date is after the date of end of last infusion + 140 days.

The selection of data for presentation by visit in these analyses is described in Table 6.7: 1.

Treatment groups for the analysis will be labelled as follows:

- "Placebo"
- "Speso 1200mg IV q4w"
- "Overall Total" (across all arms), where appropriate.

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all patients in the database (i.e., enrolled patients). Consistency check listings (for identification of violations of time windows) and a list of protocol deviations will be provided to be discussed at the RPM/DBLM/MQRM. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be queried in the clinical database. Each protocol deviation must be assessed to determine whether it is an important Protocol Deviation (iPD). For definition of iPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any iPDs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM/MQRM minutes via an accompanying Excel spreadsheet (3). The following table contains the categories which are considered to be iPDs in this trial. If the data show other iPDs, for example, based on monitor visits to the sites, then this table will be supplemented accordingly by the time of the RPM/DBLM/MQRM. Not all iPDs will lead to exclusion from analysis sets. IPDs leading to exclusion from analysis sets are indicated as such in Table 6.2: 1.

IPDs will be summarised and listed for the randomized set.

Table 6.2: 1 Handling of iPDs

| Catego | orv / | | | |
|---|---|---|---|---|
| Code | J | Description | Comments | Excluded from <sup>1</sup> |
| A | | Entrance criteria violated | | |
| <b>A1</b> | | Inclusion criteria not met | | |
| | A1.01 | 18-75 years, males or females (at Visit 1 | IC01 | None |
| | | and 2) | Also check versus derived | |
| | | LABEL: | age for patient. | |
| | | Age beyond 18-75. | | |
| | A1.02 | Body weight ≤120 kg (at Visit 1 and 2) | IC02 | None |
| | | <u>LABEL:</u> | Also check versus reported | |
| | | Weight beyond 120kg. | body weight for patient | |
| | A1.03 | Diagnosis of ulcerative colitis ≥5 months | IC03 | None |
| | | prior to screening by clinical and | Also check derived time | |
| | | endoscopic evidence and corroborated | since diagnosis for patient | |
| | | by a histopathology report. | | |
| | | LABEL: | | |
| | | Diagnosis too recent / insufficiently | | |
| | 4 1 0 4 | documented. | 1004 | DDG |
| | A1.04 | Receiving their TNFi treatment with | IC04 | PPS |
| | | infliximab (INF) with doses unchanged | | |
| | | for ≥4 months prior to randomisation and detectable drug trough levels in | | |
| | | blood; or adalimumab or golimumab | | |
| | | with doses unchanged for ≥2 months | | |
| | | prior to randomisation and detectable | | |
| | | drug trough levels in blood | | |
| | | LABEL: | | |
| | | TNFi treatment changed / not detectable. | | |
| | A1.05 | Mild or moderate disease activity, | IC05 | PPS |
| | | defined as: | Also check derived total | |
| | | Total Mayo Score (MCS) (≤10), with | MCS and mESS at baseline, | |
| | | - modified endoscopic subscore | and distance from anal verge | |
| | | $(mESS) \ge 2$ , AND | at baseline | |
| | | - disease extending 5 cm or more | | |
| | | from anal verge | | |
| | | <u>LABEL:</u> | | |
| | | Disease activity not mild or moderate. | | |
| | A1.06 | If patients receive concurrent UC | IC06 | |
| | | treatments, these need to be on stable | Also manually review | PPS |
| | | doses. | concomitant medications as | |
| | | LABEL: | use of concurrent UC | |
| | | UC treatment not on stable dose. | treatment. | |
| | | | If patients receive unstable | |
| | | | dose of probiotics, they will | |
| | | | not be excluded from PPS | |

Table 6.2: 1 (cont'd) Handling of iPDs

| Category<br>Code | ory / | Description | Comments | Excluded from <sup>1</sup> |
|---|---|---|---|---|
| Code | A1.07 | Patients with extensive colitis of >10 | IC07 | None Excluded from |
| | | years duration or family history of | | |
| | | colorectal cancer or personal history of | | |
| | | increased colorectal cancer risk must | | |
| | | have had an negative colorectal cancer | | |
| | | screening within <1 year prior to | | |
| | | screening (otherwise to be done during | | |
| | | screening colonoscopy). <u>LABEL:</u> | | |
| | | Increased risk for colorectal cancer | | |
| | A1.08 | Women of childbearing potential | IC08 | None |
| | 711.00 | (WOCBP) and men able to father a child | 1000 | Tione |
| | | must use highly effective methods of | | |
| | | birth control per ICH M3 (R2) that result | | |
| | | in a low failure rate of less than 1% per | | |
| | | year when used consistently and | | |
| | | correctly. | | |
| | | <u>LABEL:</u> | | |
| | | Contraception methods not used. | | |
| 12 | | Exclusion Criteria | | |
| | A2.01 | Extensive colonic resection, subtotal or | EC01 | None |
| | | total colectomy | | |
| | | LABEL: | | |
| | 4 2 02 | Extensive resection, or colectomy. | F.C.0.2 | N.T. |
| | A2.02 | Ileostomy, colostomy, or known fixed | EC02 | None |
| | | symptomatic stenosis of the intestine | | |
| | | <u>LABEL:</u> Ileostomy, colostomy, or stenosis. | | |
| | A2.03 | Prior use of more than two different | EC03 | PPS |
| | A2.03 | TNF inhibitor or vedolizumab | Also check the historical | 115 |
| | | LABEL: | medication | |
| | | Use of more than two different TNF | medication | |
| | | inhibitors or vedolizumab. | | |
| | A2.04 | Any treatment limiting safety or | EC04 | PPS |
| | | tolerability issue of the concurrent TNF | | |
| | | inhibitor | | |
| | | <u>LABEL:</u> | | |
| | | Treatment limiting issue of TNFi. | | |
| | A2.05 | Concurrent treatment with rectal 5-ASA | EC05 | PPS |
| | | compounds, parenteral or rectal | | |
| | | corticosteroids (incl. budesonide) within | | |
| | | 2 weeks, any investigational drug within | | |
| | | 12 weeks or 5 half-lives, whatever is | | |
| | | longer, or any prior dose of natalizumab | | |
| | | or rituximab prior to screening | | |
| | | LABEL: | | |
| | | Co-treatment not as allowed. | | |

Table 6.2: 1 (cont'd) Handling of iPDs

| Categ | ory / | | | |
|---|---|---|---|---|
| Code | 3 | Description | Comments | Excluded from <sup>1</sup> |
| | A2.06 | Patients who must or wish to continue the intake of restricted medications (see CTP Section 4.2.2.1) or any drug considered likely to interfere with the safe conduct of the trial <a href="LABEL:">LABEL:</a> Use of restricted medication. | EC06 | PPS |
| | A2.07 | Evidence of infection with C. difficile or other intestinal pathogen <28 days prior to screening LABEL: Infection with intestinal pathogen. | EC07 | PPS |
| | A2.08 | Currently require or are anticipated to require surgical intervention for UC LABEL: Requires surgical intervention for UC. | EC08 | PPS |
| | A2.09 | Colonic moderate or severe mucosal dysplasia LABEL: Colonic mucosal dysplasia. | EC09 | None |
| | A2.10 | Colonic adenomas (unless properly removed) LABEL: Colonic adenomas. | EC10 | None |
| | A2.11 | Primary sclerosing cholangitis <u>LABEL:</u> Primary sclerosing cholangitis. | EC11 | None |
| A3 | A2.12 | Faecal transplant ≤6 months before screening <u>LABEL</u> : Faecal transplant within 6 months. <i>Infectious Disease Exclusion Criteria</i> | EC12 | None |
| | A3.01 | Increased risk of infectious complications (e.g. recent pyogenic infection, any congenital or acquired immunodeficiency (e.g. HIV), live vaccination within 6 weeks prior to screening, past organ or stem cell transplantation) LABEL: Increased risk of infectious complications. | EC13 | None |
| | A3.02 | Active or latent TB (Patients with positive QuantiFERON TB test are excluded. Patients with suspected false positive or undeterminable QuantiFERON TB result may be retested) LABEL: Active or latent TB. | EC14 | None |

Table 6.2: 1 (cont'd) Handling of iPDs

| Categ | gory / | | | |
|---|---|---|---|---|
| Code | • | Description | Comments | Excluded from <sup>1</sup> |
| <b>A</b> 4 | A3.03 | Any severe infection <30 days prior to screening, including chronic or acute hepatitis B or C infection <a href="LABEL:">LABEL:</a> Severe infection within 30 days. General Exclusion Criteria | EC15 | None |
| A4 | A4.01 | Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin <a href="LABEL:">LABEL:</a> Malignancy within last 5 years. | EC16 | None |
| | A4.02 | Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomisation or planned during the study, e.g. hip replacement. LABEL: Recent or planned major surgery. | EC17 | None |
| | A4.03 | Pathological safety lab parameters: haemoglobin <8.5 g/dL, total white blood count (WBC) <3500 cells/μl, neutrophils <1000 cells/μl, thrombocytes <75.000/μl, albumin <30 g/l, creatinine ≥2 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x ULN, total bilirubin >1.5 x ULN (patients with Gilbert's syndrome are not excluded). LABEL: Pathological safety lab parameters abnormal. | EC18 Also check corresponding safety lab parameters at baseline | None |
| | A4.04 | Currently enrolled in another investigational device or drug study, or less than 12 weeks (or 5 half-lives, whichever is greater) since ending another investigational device or drug study(s), or receiving other investigational treatment(s) LABEL: Recent enrollment in other study. | EC19 | None |
| | A4.05 | Women who are pregnant, nursing, or who plan to become pregnant while in the trial LABEL: Pregnant or nursing. | EC20 | None |

Table 6.2: 1 (cont'd) Handling of iPDs

| Categ<br>Code | | Description | Co | mments | Excluded fi | rom <sup>1</sup> |
|---|---|---|---|---|---|---|
| | A4.06 | Evidence of a current | or previous EC | | None | |
| | | disease, medical cond | lition (including | | | |
| | | chronic alcohol or dru | ig abuse) other | | | |
| | | than ulcerative colitis | , surgical | | | |
| | | procedure, medical ex | | | | |
| | | (including vital signs | and | | | |
| | | electrocardiogram (E | | | | |
| | | value at the screening | | | | |
| | | reference range that in | | | | |
| | | investigator is clinica | | | | |
| | | would make the study | | | | |
| | | unreliable to adhere to | | | | |
| | | complete the trial, con | | | | |
| | | safety of the patient, | | | | |
| | | quality of the data | 1 | | | |
| | | LABÉL: | | | | |
| | | Unreliable protocol a | dherence or | | | |
| | | compromised safety. | | | | |
| 3 | | Informed consent | | | | |
| | B.01 | | | nent, not simply the tick | All | # |
| | | not available | box | , 1 3 | analyses | |
| | | LABEL: | Date of informed conser | nt missing or no | | |
| | | IC not available. | | Declaration of Informed | | |
| | | TO HOU WY WHAT HOLD. | Consent" | or informed | | |
| | | | | ata will not be used at all. | | |
| | B.02 | Informed consent | Informed consent date v | | None | |
| | 2.02 | too late | | , we wrote 1 and 1 | 1,0110 | |
| | | LABEL: | | | | |
| | | IC too late. | | | | |
| 7 | | Trial medication | | | | |
| _ | | and | | | | |
| | | randomisation | | | | |
| C1 | | Incorrect trial | | | | |
| / <b>1</b> | | medication | | | | |
| | C1.01 | Incorrect | Placeho natient who rec | eived >= 1 vial (150mg) | PPS | |
| | C1.01 | medication received | | verall /at any dosing visit | 115 | |
| | | by patients in | Can only be finally judg | | | |
| | | placebo arm | unblinding information | | | |
| | C1.02 | Incorrect | BI patient who received | | PPS | |
| | C1.02 | medication received | treatment that was rando | _ | 110 | |
| | | by patients in BI | considered an iPD. | omized would be | | |
| | | arm | Patients randomized to | RI 655130 1200mg | | |
| | | ailli | q4w, but received any > | | | |
| | | | - | · • | | |
| | | | 655130 verum different | from planned at any | | |
| | | | visit or overall | and after interior DDI | | |
| | | | Can only be finally judg | | | |
| | | | since unblinding inform | lation is required | | |

Table 6.2: 1 (cont'd) Handling of iPDs

| Categ | - | | | Excluded | |
|---|---|---|---|---|---|
| Code | | Description | Comments | from <sup>1</sup> | |
| C2 C2.01 | | Non-compliance Non-compliance with study drug intake administered dose too low | Administered overall infusion volume is less than 80% of the total planned volume. The total planned volume is | PPS | |
| | C2.02 | Non-compliance with study drug intake administered dose too high | <ul> <li>60mL if discontinuation up to and including visit V2</li> <li>120mL if discontinuation up to and including V4</li> <li>180mL if discontinuation up to and including V5</li> <li>The total planned volume overall is 180 mL.</li> <li>Administered overall infusion volume is greater than 120% of the total planned volume</li> <li>The total planned volume is</li> <li>60mL if discontinuation up to and including visit V2</li> <li>120mL if discontinuation up to and including V4</li> <li>180mL if discontinuation up to and including V5</li> <li>The total planned volume overall is 180 mL.</li> </ul> | None | |
| C3 | C3.01 | Randomization not followed Treated without randomisation LABEL: Treated without randomisation. | Patient treated according to eCRF, but not randomised according to IVRS. | RS(i),<br>SAF(i),<br>FAS(i),<br>PPS | |
| <b>C4</b> | | Medication code broken | | | |
| | C4.01 | Medication code broken inappropriately <a href="LABEL">LABEL</a> : Medication code broken inappropriately | Medication code was broken prior to Week 12 for no valid reason. Final decision at the DBL meeting for the Week 12 analysis based on medical judgment. | PPS | # |
| D | | Concomitant medication | | | |
| D1 | D1.01 | Previous medication Washout of previous medication too short LABEL: | | PPS | # |
| D2 | D2.01 | Washout too short. Prohibited medication use Use of restricted medication as per CTP Table 4.2.2.1: 1 during the on-treatment period when not provided as a rescue treatment to stabilize a worsening disease condition – prior to or up to Week 12 | | PPS | # |
| | | LABEL: Restricted medication prior to Week 12 | | | |

Table 6.2: 1 (cont'd) Handling of iPDs

| Categ | ory / | | | | |
|---|---|---|---|---|---|
| Code | | Description | Comments | Excluded from <sup>1</sup> | |
| | D2.02 | Use of restricted medication as per CTP Table 4.2.2: 1 when not provided as a rescue treatment to stabilize a worsening disease condition - after Week 12 LABEL: Restricted medication after Week 12 | | None | # |
| D3 | | Change in Background medication | Note: Background<br>medication is split into:<br>• concurrent UC treatments<br>• Background TNFi medi-<br>cation (e.g. infliximab) | | |
| | D3.01 | Concurrent UC treatments need to be on stable doses prior or up to Week 12: Oral 5-ASA compounds <u>LABEL:</u> Oral 5-ASA compounds not stable | Medical review, per investigator's judgement, any dose increase used as rescue treatment due to disease worsening or not improved, this will not be considered as iPD. Only dose increase not as rescue use will lead to exclusion from PPS | PPS | # |
| | D3.02 | Concurrent UC treatments need to be on stable doses prior or up to Week 12: Oral corticosteroids LABEL: Oral corticosteroids not stable | Medical review, per investigator's judgement, any dose increase used as rescue treatment due to disease worsening or not improved, this will not be considered as iPD. Only dose increase not as rescue use will lead to exclusion from PPS | | # |
| | D3.03 | Concurrent UC treatments need to be on stable doses prior or up to Week 12: Azathioprine, 6-mercaptopurin or methotrexate LABEL: Azathioprine 6-mercaptopurin or methotrexate not stable | Medical review, per investigator's judgement, any dose increase used as rescue treatment due to disease worsening or not improved, this will not be considered as iPD. Only dose increase not as rescue use will lead to exclusion from PPS | PPS | # |

Table 6.2: 1 (cont'd) Handling of iPDs

Trial No: 1368-0010 - 3.0 (Final)

| Categ | ory / | | | | |
|---|---|---|---|---|---|
| Code | | Description | | Excluded from <sup>1</sup> | |
| | D3.04 | Concurrent UC treatments need to be on stable doses prior or up to Week 12: Probiotics (e.g. S. boulardii) LABEL: Probiotics not stable | Medical review | None | # |
| | D3.05 | Any dose change in background TNF inhibitor medication when not provided as a rescue treatment to stabilize a worsening disease condition – prior to or up to Week 12 <u>LABEL</u> : Dose change in background TNFi prior Week 12 | Dose change in background<br>TNF inhibitor therapy is<br>not allowed per CTP<br>section 4.2.2 from<br>Screening through End of<br>Treatment. | i PPS | # |
| | D3.06 | Any dose change in background TNF inhibitor medication when not provided as a rescue treatment to stabilize a worsening disease condition – after Week 12 <u>LABEL</u> : Dose change in background TNFi after Week 12 | Dose change in background<br>TNF inhibitor therapy is<br>not allowed per CTP<br>section from Screening<br>through End of Treatment. | None | # |
| E | | Missing data | <not specified=""></not> | | |
| F | | Study specific analysis | <not specified=""></not> | | |
| F1 | | Other trial specific violation | <not specified=""></not> | | |
| | F1.01 | Incomplete diagnosis of ulcerative colitis<br>LABEL: | Medical review | PPS | # |
| | F1.02 | Incomplete diagnosis of UC Primary endpoint assessment more than 2 weeks before planned day LABEL: Primary endpoint assessment > 2 weeks before planned. | | PPS | |
| F2 | | Certain violations of procedures used to measure primary or secondary efficacy data | <not specified=""></not> | | |
| G | G1 | Other safety related violations Pregnancy test not done for woman of child bearing potential or pregnant during study LABEL: Pregnancy test not done | Pregnancy test not done at<br>any visit where such is<br>scheduled | None | |

<sup>#</sup> PV will be detected manually

Source: BI reference document: "Identify and Manage Important Protocol Deviations (iPD)" [ 001-MCS-40-413] (2).

<sup>&</sup>lt;sup>1</sup>For specification on definition of analysis sets, refer to <u>Section 6.3</u>. Analysis of efficacy data according to the PPS will not be done at the time of the 1<sup>st</sup> interim database snapshot.

### 6.3 SUBJECT SETS ANALYSED

The following analysis sets will be defined for this trial:

- Enrolled set (ES):
  - This patient set includes all patients who signed the informed consent form. It will be used for analyses of patient disposition.
- Randomized set (RS):
  - This patient set includes all patients who were randomized into the trial. It will be used for analyses of patient disposition and patients with iPDs.
- Safety analysis set (SAF):
  - This patient set includes all randomized patients who received at least one dose of study drug. It will be the main analysis set for presentation of safety. Treatment assignment will be analyzed according to the actual treatment.

For the primary analysis to be performed once all patients have completed through the Week 12 visit, and the final trial analysis, the following additional patient sets will be defined.

- Full analysis set (FAS):
  - This patient set includes all patients in the SAF who had a baseline measurement available for the primary endpoint. Treatment assignment will be as randomized. This is the main analysis set for presentation of efficacy.
- Per protocol set (PPS):
  - This patient set includes all patients in the FAS who adhered to the CTP without any iPDs which are flagged for exclusion from the PPS in the table above. This set will be used for sensitivity analysis on the primary efficacy endpoint.

For the first interim database snapshot, modified versions of the ES, RS, SAF, and FAS will be defined: the ESi, RSi, SAFi, and the FASi. Each of the modified patient sets will include those patients from the original set who completed/discontinued through the Week 12 visit on or prior to the cut-off date (see <u>Section 3</u>). Each of these modified patient sets will be handled according to the same procedures used to derive the full patient sets.

For the analyses to be performed at the time of the second interim database snapshot (when all randomized patients have completed/discontinued through Week 12), the ES, RS, SAF, FAS, and PPS will be used. Corresponding analyses performed at the time of the first interim database snapshot will use the ESi, RSi, SAFi, and FASi.

For the final analysis, the ES, RS, SAF, FAS, and PPS will be used.

The discussion of all exceptional cases and problems and the decisions on the allocation of patients to populations will be made at latest at the DBLM. A separate DBLM will be held prior to each database snapshot of this trial.

### **Handling of Treatment Misallocations in Analysis Sets**

If a subject is randomized but not treated, by definition such patients are excluded from FAS and PPS for efficacy analysis and excluded from SAF for safety analyses as no study medication was taken. However, they will be included in RS and reported under their randomized treatment group for sensitivity efficacy analysis. Please refer to Section 7.4 for more details.

If a subject is treated but not randomized, they will be excluded from both efficacy analysis and safety analysis by definition. However, subjects under such circumstances will be summarized in the final clinical trial report.

If a subject is randomized but took incorrect treatment during the study, then:

- For efficacy analyses according to FAS, PPS, and RS, they will be reported under their randomized treatment groups. But if the subject has an iPD as defined in Section 6.2, then they will be excluded from PPS for efficacy analysis.
- For safety analyses using the SAF,
  - if a subject is randomized with BI 655130 1200mg q4w treatment, then they will be reported under their randomized treatment group for safety analysis because the overall safety profile will be driven by the amount of drug received in totality over the entire treatment duration. It is not likely that the safety profile will deviate from the planned treatment regimen if the subject receives only one or two vials of the incorrect medication during only some dosing occasions. The subject will be assigned to the placebo treatment group only if they don't receive any BI 655130 during the entire treatment period.
  - if a subject is planned with placebo treatment group, then they will be reported under placebo if no treatment with BI 655130 is received at any visit. If the subject receives > = 1 vial (> = 150mg) of BI 655130 during the entire treatment duration, then they will be reported as BI 655130 1200mg treatment group.

<u>Table 6.3: 1 (first interim database snapshot)</u>, and <u>Table 6.3: 2</u> (second interim database snapshot and final trial snapshot) illustrate the data sets which will be used for each category class of endpoints, and the approaches used with regard to missing data. For explanation of the different methods of handling missing data see <u>Section 6.6</u>.

Trial No: 1368-0010 - 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 1 Subject sets analysed (first interim database snapshot)

| Patient set | | | | |
|---|---|---|---|---|
| Class of endpoint | RSi | ESi | SAFi | FASi |
| Disposition | | OR | | OR |
| Compliance | | | | OR |
| Exposure | | | OR | |
| iPDs | OR | | | |
| Demographic/baseline characteristics | | | | OR |
| Primary endpoint | NRI*, OC* | | | NRI,<br>OC |
| Secondary efficacy endpoints | NRI*, OC* | | | NRI,<br>OC |
| Further efficacy endpoints | | | | All: OC<br>Binary: NRI<br>Continuous: MMRM |
| PK concentr.& ADA&DNA | | | OC (if available) | |
| Biomarker endpoints | | | OC (CRP, FLF,<br>FCP. Others: if<br>available) | |
| Safety parameters | | | OR,<br>OC-IR | |
| Use of rescue medication | | | | OR |

For explanation of the different approaches with regard to missing data see Section 6.6.

At the time of the first interim database snapshot, only the primary analysis on each efficacy endpoint will be done. All safety displays will be produced. No inferential subgroup analyses will be performed.

OR = original results.

 $NRI = No \ Response \ Imputation \ excluding \ values \ after \ rescue \ medication \ taken$ 

OC = observed cases excluding values after rescue medication taken

OC-IR = observed cases including also values after rescue medication taken

LOCF = Last observation carried forward

<sup>\*</sup>only when RS are different from FAS

Trial No: 1368-0010 - 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 2 Subject sets analysed (second interim database snapshot and final trial snapshot)

| | | | Patient se | t | |
|---|---|---|---|---|---|
| Class of endpoint | RS | ES | SAF | FAS | PPS |
| Disposition | | OR | | OR | |
| Compliance | | | | OR | |
| Exposure | | | OR | | |
| iPDs* | OR | | | | |
| Demographic/baseline characteristics | | | | OR | |
| Primary endpoint | NRI**, OC** | | | NRI,<br>OC | NRI,<br>OC |
| Secondary efficacy endpoints | NRI**, OC** | | | NRI,<br>OC | |
| Further efficacy endpoints | | | | All: OC<br>Binary: NRI<br>Continuous: MMRM | |
| PK concentr.& ADA&DNA | | | OC | | |
| Biomarker endpoints | | | OC | | |
| Safety parameters | | | OR,<br>OC-IR | | |
| Use of rescue medication | | | | OR | |

For explanation of the different approaches with regard to missing data see Section 6.6.

At the time of the second interim and final trial database snapshots, all analyses per TSAP are scheduled to be performed.

 $OR = \hat{original}$  results.

NRI = No Response Imputation excluding values after rescue medication taken

OC = observed cases excluding values after rescue medication taken

OC-IR = observed cases including also values after rescue medication taken

LOCF = Last observation carried forward

<sup>\*</sup> any patient with the iPD of treated but not randomized (C3.02) will only be listed in the footnote of the iPD table.

<sup>\*\*</sup>only when RS are different from FAS



#### 6.5 POOLING OF CENTRES

Given the low number of patients per centre and the primarily descriptive nature of the statistical analysis, separate analyses by centre are not meaningful and not desirable. All patients from all centres will be pooled for statistical analysis.

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Section 7.5 of the CTP describes the handling of missing data.

The original results (OR) approach implies the presentation of data exactly as observed, i.e., not using time windows and not setting values to missing.

OR analysis will be performed on parameters and endpoints that are either not affected by patients' rescue medication use (e.g., plasma concentration level of BI 655130, or rescue medication use itself), or, if it is not meaningful to apply any imputation rule for the replacement of missing values.

#### 6.6.1 Withdrawals

The reasons for withdrawal from treatment will be reported as indicated on the eCRF.

### 6.6.2 Efficacy data

Based on the different reasons for a subject to have missing data, various approaches will be used to assess the impact of missing data on the different efficacy endpoints of this trial. The approaches to be applied are described below.

Missing data imputations at the primary analysis at Week 12, that is, once all patients have achieved the Week 12 visit, will be performed using all available on-treatment data observed up to the respective analysis cut-off date.

### Binary efficacy endpoints

For all binary endpoints (i.e. endpoints that are either 1 (patient responded) or 0 (patient did not respond)), the following will be performed as the primary imputation approach (analysis type: Non Response Imputation [NRI]):

- 1. If there are data at visits both before and after the visit with a missing outcome, then impute as success only if both neighbouring visits also represent a success (independent of whether the preceding and following observations were selected for analysis based on time windows described in <u>Section 6.7</u>);
- 2. Otherwise, impute as a failure to achieve a response

If a patient takes a rescue medication as defined in <u>Section 5.4.5</u> for the treatment of ulcerative colitis prior to observing the primary endpoint for this trial, then all data subsequent to rescue treatment will be considered to represent a failure to achieve a response.

Further approaches to the handling of missing data will be performed as follows:

- Observed cases (analysis type: OC) approach will be used as a sensitivity analysis and will include all collected data, with no imputation performed on the missing data. Such an OC approach will exclude all values measured after intake of a rescue medication (i.e. such values will be set to missing).
- Observed cases including rescue (analysis type: OC-IR) approach will be used as a further sensitivity analysis and is an extension of the OC approach which includes all values which were measured after rescue medication intake.

Missing data after premature discontinuation will not be imputed when following the OC and OC-IR approach.

## Continuous further efficacy endpoints

For further efficacy endpoints which are continuous in nature, the use of a restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach, if applicable, will ensure that missing data are handled implicitly, via a missing at random assumption, by the statistical model.

The continuous further efficacy endpoints will also be summarized by visits descriptively via the OC approach (described above for the binary efficacy endpoints).

### 6.6.3 Safety data

**From CTP Section 7.5**: With respect to safety evaluations, it is not planned to impute missing values.

For safety data that are displayed by time point (or visit) of measurement, the OC-IR approach will be used.

The only exceptions where imputation might be necessary for safety evaluation are AE dates and start and stop dates for concomitant medications. Missing or incomplete AE dates are imputed according to BI standards (see *BI-KMED-BDS-HTG-0035*: "Handling of missing and incomplete AE dates" (4)).

Partial start and stop dates for concomitant medications and background, rescue, as well as historical medication for UC will be imputed to enable subsequent calculation (but not for display) by the following "worst case" approach:

- If the day of the end date is missing, then the end date is set to last day of the month (or to the patient's trial completion date, if it is earlier than the last day of the month).
- If the day and month of the end date are missing then the end date is set to 31st of December of that year (or to the patient's trial completion date, if it is earlier than the 31st of December of that year).
- If the day of the start date is missing the start date is set to the first day of the month (except for rescue medication, where the first dosing day will be used if first dosing happened in the same month).
- If the day and month of the start date are missing then the start date is set to the 1<sup>st</sup> of January of that year (except for rescue medication, where the first dosing day/month will be used if the first dosing happened in the same year).

All other cases need to be assessed by the trial team on an individual basis, using the above points as guidance.

#### 6.6.4 **PK data**

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472 RD-01) (5).

### 6.6.5 **Biomarker data**

Missing biomarker data (NOS - no sample, NOR - no valid result, NOA - not analysed) will not be imputed.

Trial No: 1368-0010 - 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For disease specific (protein) markers (from serum or stool samples) the following handling of data below or above the limit of quantification will be applied:

- BLQ data will be replaced by 0.5 · LLOQ. Hereby LLOQ will be the maximum used lower reference limit for classification of BLQs. All values lower than LLOQ will be imputed (regardless of whether they are classified as BLQ or not).
- ALQ data will be replaced by ULOQ, if ULOQs are available and are greater than observed study values (i.e. the highest solution was applied for the measurement). Otherwise, ALQ data will be excluded from the analysis.

The OC approach (see Section 6.6.2) will be used to present the data.

The handling of other biomarkers, e.g. RNA expression, will be specified in a separate document.

### 6.6.6 Time since first diagnosis

For incomplete information on the date of first diagnosis, time since first diagnosis will be calculated as follows:

- If the year of first diagnosis is unknown, then time since first diagnosis will be set to missing.
- If day and month of the first diagnosis are unknown, then time since first diagnosis will be calculated as if diagnosed on the 30<sup>th</sup> of June of that year.
- If only the day of the first diagnosis is unknown, then time since first diagnosis will be calculated as if diagnosed on the 15<sup>th</sup> of that month.

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Measurements reported with the date and time and that were taken prior to start of administration of trial treatment will be considered pre-treatment values. Measurements reported with a date only (and no time) and that were taken on the day of first administration of trial treatment will also be considered pre-treatment values. These pre-treatment values will be assigned to visits according to the nominal visit number as recorded on the eCRF, or as provided by the laboratory.

Baseline, unless otherwise specified, is defined as the last measurement collected prior to the start of administration of the trial treatment.

Measurements taken after the start of administration of the trial treatment will be considered either on- or off-treatment values based on the definition in <u>Section 6.1</u>, and will be assigned to visits for statistical analysis, if applicable, as defined in <u>Table 6.7: 1</u>.

Neither analysis of AE data, concomitant medication, non-drug therapies, nor use of rescue medication will be based on visits. Therefore, no assignment to time windows will be necessary.

Frequency tables for AE data will be using on-treatment data only up to the time of the planned trial analysis (Week 12, or Week 36). Frequency tables for concomitant medication, non-drug therapies, and rescue medication will be based on all available data up to the time

of the planned trial analysis (Week 12, or Week 36).

For derivation of the last value on treatment, minimum value on treatment, and maximum value on treatment, all on-treatment values (whether or not selected in any time window; see Table 6.1: 1 for definition of the on-treatment period) will be considered; these will be derived for analysis of laboratory and vital signs data. For identification of potentially clinically significant abnormal laboratory values, all values (whether or not selected in any time window) before the off-treatment period will be considered.

A graphical analysis of the ALT and total bilirubin will be performed (so called eDISH plot) based on the available data obtained during the on-treatment period.

All other safety, efficacy, and biomarker measurements will be assigned to visits based on extended time windows around the planned visit dates defined relative to the day of first trial treatment (which is scheduled for Visit V2). These extended time windows are defined in Table 6.7: 1.

Table 6.7: 1 Time windows for assignment of efficacy, safety lab, vital signs and biomarker to visits for statistical analysis

| Visit | | Planned | | Tiı | me window (I | Days) | |
|---|---|---|---|---|---|---|---|
| number | Visit label | day | Window | Start | End | Start | End |
| /name | | | (per CTP) | (per CTP) | (per CTP) | (extended) | (extended) |
| V1a | Screening | -35 to -8 | n/a | | | | |
| Vlb | Screening | - 28 to -6 | n/a | | | | |
| V2 | Baseline | Day 1 | +/- 0 | 1 <sup>A</sup> | 1 <sup>A</sup> | ≤1 <sup>A</sup> | 1 <sup>A</sup> |
| On-treatr | nent data only | | | | | | |
| V3 | Week 2 | Day 15 | +/- 2 | 13 | 17 | 2 | 22 |
| V4 | Week 4 | Day 29 | +/- 3 | 26 | 32 | 23 | 43 |
| V5 | Week 8 | Day 57 | +/- 3 | 54 | 60 | 44 | 71 |
| EOT | Week 12/EoT | Day 85 | +/- 4 | 81 | 89 | 72 | 99* |
| FU1 | Week 16/FU1 | Day 113 | +/- 4 | 109 | 117 | 100 | 134 |
| FU2 | Week 22/FU2 | Day 155 | +/- 4 | 151 | 159 | 135 | Min(175, |
| | | | | | | | LD+140) |
| | on- and off-treatn | nent) | | | | | |
| FU3 <sup>B</sup> | Week 28/FU3 | Day 197 | +/- 4 | 193 | 201 | 176 | 225 |
| EOS B | Week 36/EOS | Day 253 | +/- 4 | 249 | 257 | 226 | Day of last |
| | | - | | | | | follow up |
| | | | | | | | value <sup>B</sup> |

For primary analysis for efficacy (Week 12) – Data after minimum (cut-off<sup>C</sup>, Day 99) will not be used for analyses

For final analysis – Data after (LD<sup>D</sup> + 140) will not be used for any planned on-treatment analyses

Days are counted relative to the day of first treatment, which is defined as Day 1.

A Note that measurements made at Day 1 and assigned to the on-treatment period (because mistakenly made after start of infusion of trial treatment) via assessment on date and time (i.e. safety laboratory) will not be assigned to Day 1. Such data will be listed only.

<sup>&</sup>lt;sup>B</sup> Note that measurements assigned to the Week 28/FU3 or Week 36/EOS visits but after LD+140 are intended to represent off-treatment (i.e., follow-up) measurements, as they are made after the end of the on-treatment
# period.

<sup>©</sup> The cut-off date is not applicable for the final trial analysis.

Repeated and unscheduled efficacy, safety, and biomarker measurements will be handled similarly to scheduled measurements and will also be assigned to a time window depending upon the date of measurement.

Only one observation per time window will be selected for statistical analysis at a particular visit – the value which is closest to the protocol planned visit day will be selected. If there are two observations which have the same difference in days to the planned day, the later value will be selected. If there are two observations on the same day, then for vital signs the latest value (according to the date and time) will be selected, and for other endpoints the worst value will be selected.

Assignment of efficacy observations to visits based on time windows will be based on the non-imputed (observed) data after setting values after rescue medication intake to missing (if applicable, i.e. for the "NRI" and the "OC" approaches defined in Section 6.6).

For visits without an assigned value based on time windows, a value will thereafter be imputed as defined in <u>Section 6.6</u>. Imputation of efficacy endpoints, when applicable, will be performed based on all available observations obtained, irrespective of whether the observation was selected in any time window.

D LD = Day of Last dose/infusion received

# 7. PLANNED ANALYSIS

All efficacy analyses will be purely exploratory in nature. The following analyses are planned at different stages throughout the trial.

# • First Interim Database Snapshot – Week 12 Analysis

The analysis will be performed using all randomized patients who completed/discontinued through the Week 12 visit on or prior to the cut-off date (see Section 3). A database snapshot will then be done. At this time, an interim analysis of the efficacy and safety data through Week 12 will be performed by the sponsor.

The individual patient cut-off date for inclusion of data into the analysis is the minimum of the analysis-specific cut-off date, or study day 99, as described in Table 6.7: 1.

The analyses for this snapshot will be performed using the subject sets of ESi, RSi, SAFi, and FASi (see Section 6.3).

#### • Second Interim Database Snapshot – Week 12 Analysis (Primary Analysis for CTR)

The analysis will be performed using all randomized patients who completed/discontinued through the Week 12 visit. A database snapshot will then be done. At this time, a complete analysis of all efficacy, safety, and PK/Biomarker data will be done through Week 12, and will be performed by the sponsor.

The individual patient cut-off date for inclusion of data into the analysis is the minimum of the analysis-specific data cut-off, or study day 99, as described in <u>Table 6.7: 1</u>.

The analyses as described in <u>Section 6.3</u> of this TSAP will be performed using the subject sets of ES, RS, SAF, FAS, and PPS.

# • Final analysis (Week 36)

The analyses of the entire efficacy, safety, and biomarker data collected through the full 36 weeks of follow-up will be performed once all entered patients have completed the trial (up to EOS Visit); at that time point, a final database lock will be done and all on treatment data through Week 36 will be reported.

#### General Remarks

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (001-MCG-159) (10).

The individual values of all patients will be listed, including those collected during the off-treatment period. Listings will generally be sorted by country, centre number, patient number, and visit (if visit is applicable in the respective listing). AE listings will be sorted by treatment (see Section 7.8.1 below for details).

The following standard descriptive statistical parameters will be displayed in summary tables for continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Q1 lower quartile

Median median

Q3 upper quartile Max maximum

Statistical parameters will be displayed to a defined number of decimal places as specified in the BI guideline "Reporting of Clinical Trials and Project Summaries" (10).

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group; unless otherwise specified, this includes all patients in the respective patient set whether they have non-missing values or not. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there are missing values.

For the final trial analysis up to Week 36, displays of certain safety endpoints, such as AE, will be produced only for the on-treatment period. Displays of endpoints presented by-visit, additional outputs, which include both on- and off-treatment data, will be produced at the time of update analysis after final DBL (see also Section 6.7).

Disposition of the patient population participating in the trial will be summarised by presentation of the frequency of patients screened, entered, screened but not entered, treated, entered but not treated, who completed all doses of trial medication as planned, who completed the EOT visit, who completed the EOS visit, and who were prematurely discontinued, by reason. Disposition will be listed by country.

The frequency of patients with iPDs will be presented for the RS by treatment. The iPDs will be listed per patient indicating whether or not the iPD led to exclusion from patient sets analysed.

The frequency of patients in each of the different analysis sets will also be presented by treatment.

All Section 7 analyses described below are presented for the second interim database snapshot (based on all randomized patients) and the final analysis using the subject sets of ES, RS, SAF, FAS, and PPS. A sub-selection of these analyses will be performed at the time of the first interim database snapshot using the subject sets of ESi, RSi, FASi, and SAFi.

# 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR.

Descriptive statistics will be presented by treatment for demographic parameters and baseline characteristics based on the FAS.

For the continuous variables described below, the following categories will be defined and presented according to the number and percentage of patients in each category:

Categories for summary of continuous variables Table 7.1: 1

| | ~ . |
|----------------------------|--------------------------------------|
| Variable | Categories |
| Age | < 50 years |
| | 50 to < 65 years |
| | 65 to < 75 years |
| | ≥ 75 years |
| | < 65 years |
| | ≥ 65 years |
| Weight | ≤70 kg |
| | $>70 \text{ to } \leq 80 \text{ kg}$ |
| | $>80 \text{ to} \le 90 \text{ kg}$ |
| | >90 kg |
| BMI | $< 25 \text{ kg/m}^2$ |
| | $25 \text{ to} < 30 \text{ kg/m}^2$ |
| | $\geq 30 \text{ kg/m}^2$ |
| Time since first diagnosis | ≤ 1 year |
| Time since mist diagnosis | $> 1$ to $\le 5$ years |
| | $> 5$ to $\le 10$ years |
| | > 10 years |
| Total MCS at baseline | < 4 |
| | 4 to <6 |
| | 6 to <8 |
| | 8 to <=10 |

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Analyses of concomitant diseases and medication will be based on the FAS.

Concomitant diseases will be coded according to the most recent version of MedDRA.

Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary.

Concomitant non-drug therapy will be coded according to the most recent version of MedDRA.

Concomitant diseases which are present at start of the study, as well as characteristics of the trial disease, will be descriptively summarized by treatment.

Characteristics of the trial disease, such as the disease diagnosis and the type of extraintestinal diagnoses which are present at start of the study, as well as the occurrence of any prior surgery for ulcerative colitis will be descriptively summarized by treatment. During the course of the study's on-treatment period, any changes in the pre-existing extra-intestinal diagnoses (improved or worsened) by visit (including as an overall on-treatment assessment), as well as the development of newly diagnosed extra-intestinal diagnoses will also be summarized.

A medication will be considered concomitant to treatment, if it

- is ongoing at the start of trial treatment or
- starts within the on-treatment period (see <u>Section 6.1</u> for a definition of study analysis phases).

Concomitant medication use (excluding rescue medication, historical medication for UC and background medication) will be summarised by treatment with frequency and percentage of patients by preferred name. Summaries will be presented for

- concomitant medication started any time prior to the Week 12 visit (for any patient with a missing Week 12 visit, available data will be summarized up to the end of the Week 12 time window, see <u>Table 6.7: 1</u>).
- concomitant medication started any time on or after the Week 12 visit, and prior to EoS.

The frequency and percentage of patients with historical medication for UC will be displayed, and by reason for discontinuation. In addition, the reason for discontinuation will also be presented by type of medication.

The frequency and percentage of patients taking any background medication for UC will be tabulated by type of background therapy. Further displays regarding changes in background medication during the on-treatment period will be summarized in <u>Section 7.6.4</u>.

Use of rescue medication will be summarised separately (see Section 7.6.4).

Concomitant use of non-drug therapies will be summarised with frequency and percentage. Summaries will be presented for:

- concomitant non-drug therapy started any time prior to the Week 12 visit (for any patient with a missing Week 12 visit, available data will be summarized up to the end of the Week 12 time window, see Table 6.7: 1).
- concomitant non-drug therapy started any time on or after the Week 12 visit, and prior to EoS.

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will be summarised overall and by visit via total volume infused (as a % of planned) for the FAS using descriptive statistics (N, mean, SD, minimum, median, and maximum). The volume infused (as a % of planned) is defined as the volume infused at a visit (in ml as recorded in the eCRF), divided by 60 ml (the volume the patient should have received), times 100.

For the patients who discontinued the study treatment prematurely, only the visits on or before premature discontinuation will be used for the calculation of overall compliance.

The number and percentage of patients with the following overall compliance categories will be presented:

- "<50% of planned",
- "50 to <80% of planned"
- "80 to 100% of planned".

The number of patients who received a dose will be tabulated per visit.

#### 7.4 PRIMARY ENDPOINT

The binary primary efficacy endpoint will be described using patient frequencies and percentages for the FAS (or its derivatives - see <u>Section 6.3</u>). The underlying mESS will be based on central reading - replacing missing values with results based on investigator assessment.

### 7.4.1 Primary analysis of the primary endpoint

The primary analysis of the primary endpoint will be based on Section 7.3.1 of the CTP.

**From CTP Section 7.3.1:** The primary analysis of the unadjusted absolute risk difference versus placebo will be calculated simply as the difference in the observed proportion of patients with mucosal healing at Week 12, for the FAS. A 95% Newcombe confidence interval around this difference will also be provided.

The method to provide confidence intervals for single proportions will be based on the Wilson method (14). The method to provide confidence intervals for the unadjusted risk

Trial No: 1368-0010 – 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

differences is derived from the Newcombe method (15), and is constructed from the Wilson score confidence interval for each of the single proportions.

As described in Section 7.2 of the CTP, there will be no formal hypothesis testing performed in this trial.

# 7.4.2 Sensitivity analysis, subgroup analysis, exploratory analysis of the primary endpoint

The further analysis of the primary endpoint will be based on Section 7.3.1 of the CTP as below.

From CTP Section 7.3.1: Exploratory analyses of the primary endpoint will include, in the absence of model convergence issues due to occurrence of low cell frequencies, the difference in the proportion of patients with mucosal healing at Week 12 between BI 655130 and placebo, for the FAS, using a logistic regression approach with a logit link. Fixed classification effects will include treatment and presence or absence of use of infliximab (yes/no). The estimates from the logistic regression are on the logit scale, and the difference in proportions will be calculated as the difference between the predicted probabilities in the treatment groups on the original scale, with the confidence interval calculated using the cumulative distribution function method of Reeve.

Prior to the first interim database lock, it was decided that the Reeve confidence intervals will not be used due to low enrolment.

The subgroup analysis will create three logistic regression models for the primary endpoint for the covariates listed in <u>Table 6.4: 1</u>. The SAS code for the logistic regression model is as follows:

```
proc logistic data=indata;
  class trt (ref="&_j.") / param=GLM;
  model resp = trtseq &covar. / link=LOGIT CovB;
  lsmeans trt / cl ILINK;
run;
```

Other analyses of the primary endpoint will include:

- Sensitivity analyses utilizing different patients sets (such as the PPS), as well as alternative methods for the handling of missing data as described in CTP Section 7.5;
- Exploration of the relationship between various demographic or baseline characteristics data and the primary endpoint will be performed via graphical methods as well as using a logit link with

A separate logistic regression model for the primary endpoint with each of the following baseline covariates and including treatment as well as treatment-by-covariate interaction as fixed effects will be fit:

- Categorical:
  - o Sex
  - Smoking status (previous/current or never)
- Continuous:
  - o Age
  - o BMI
  - o Time to disease diagnosis

Parameter estimates from the logistic model will be presented. The estimated response rate for each treatment arm across the range of observed covariate values will be displayed graphically.

Note that exploratory and other analyses of the primary endpoint are planned to be performed at the time of the Week 12 primary analysis only, unless otherwise specified.

Table 7.4.2: 1 below summarizes the primary and further analyses as described above, together with the sensitivity analyses and subgroup analysis.

Table 7.4.2: 1 Summary of all analyses to be performed for the primary endpoint

| | Summary of analysis | | |
|---|---|---|---|
| Analysis | Analysis set | Imputation<br>Approach | Analysis model |
| Primary analysis | FAS | NRI | Unadjusted absolute risk difference |
| Sensitivity (a) -1 | RS* | NRI | Unadjusted absolute risk difference |
| Sensitivity (a) -2 | FAS | OC | Unadjusted absolute risk difference |
| Sensitivity (a) -3 | RS* | OC | Unadjusted absolute risk difference |
| Sensitivity (a) -4 | PPS | NRI | Unadjusted absolute risk difference |
| Sensitivity (a) -5 | PPS | OC | Unadjusted absolute risk difference |
| Further analysis | FAS | NRI | Adjusted risk difference via logistic regression |
| Subgroup analysis | FAS | NRI | Adjusted risk difference via logistic regression including different covariates |

Note:

For explanation of the different approaches with regard to missing data see Section 6.6.

NRI = No Response Imputation excluding data after rescue treatment

OC = Observed Cases excluding data after rescue treatment

\*Only when RS is different from FAS

Trial No: 1368-0010 – 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5 SECONDARY ENDPOINTS

# 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been specified.

7.5.1.1 Primary analysis of the key secondary endpoint(s)

This section is not applicable as no key secondary endpoints have been specified.

7.5.1.2 Sensitivity analysis, subgroup analysis, exploratory analysis of the key secondary endpoint(s)

This section is not applicable as no key secondary endpoints have been specified.

# 7.5.2 (Other) Secondary endpoints

Analysis of secondary endpoints is described in Section 7.3.2 of the CTP.

#### From CTP Section 7.3.2:

For the secondary binary endpoints, for the FAS, the unadjusted absolute risk difference versus placebo will be calculated and a 95% Newcombe confidence interval around this difference will also be provided.

A logistic regression analysis on the binary secondary efficacy endpoints, per the approach described for the primary endpoint, will also be done on the FAS. As defined for the primary endpoint, the method to provide confidence intervals for single proportions will be based on Wilson (14), and for unadjusted risk differences is derived from the Wilson method by Newcombe (15).

<u>Table 7.5.2: 1</u> below summarizes all of the analyses to be performed for the secondary endpoints.

**Trial No: 1368-0010 – 3.0 (Final)** 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.5.2: 1 Summary of all analyses to be performed for the secondary endpoints

| | Summary of analysis | | |
|---|---|---|---|
| Analysis | Analysis set | Imputation<br>Approach | Analysis model |
| Planned analysis in CTP | FAS | NRI | Unadjusted absolute risk difference |
| Sensitivity-1 | FAS | OC | Unadjusted absolute risk difference |
| Sensitivity-2 | FAS | NRI | Adjusted risk difference via logistic regression |
| Sensitivity-3* | FAS | NRI | Unadjusted absolute risk difference<br>(worst case approach on SFS/RBS<br>calculation) |

Note:

Standard approach of SFS/RBS calculation is applied unless otherwise specified.

For explanation of the different approaches with regard to missing data see Section 6.6.

NRI = No Response Imputation excluding data after rescue treatment

OC = Observed Cases excluding data after rescue treatment



<sup>\*</sup>only applicable to the secondary endpoints of clinical remission and total clinical remission and the further endpoint of clinical response.







#### 7.7 EXTENT OF EXPOSURE

The number of subjects who received a dose of trial drug will be tabulated. The duration of infusion [minutes] and the amount of treatment received [mg] (actual and weight based) will be summarised by descriptive statistics (N, mean, SD, minimum, median, maximum) per visit and overall. The total duration of exposure [days), defined as the time from start of the first infusion to time of end of the last infusion plus one day, will also be displayed.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed based on the SAF following BI standards. No hypothesis testing is planned.

For the first interim database snapshot analysis, selected safety data, such as AE listings and displays, beyond the Week 12 visit up to the earliest of the REP/cut-off date will be done for the SAFi (see Section 6.3).

For the second interim database snapshot analysis (the primary analysis for the CTR), a similar approach will be taken as above for the first snapshot. The final analysis will include all safety data up to the end of the trial.

#### 7.8.1 **Adverse events**

AEs will be coded with the most recent version of MedDRA. Patients will be analysed according to the actual treatment received.

The exposure adjusted incidence rate (per 100 subject years) of a selected treatment emergent adverse event is defined as the number of subjects experiencing the adverse event per treatment group during time at risk divided by the total time of subjects at risk in that treatment group to contribute the event to the analysis multiplied by 100 (per 100 subject years), where:

Time at risk [subject years] = (date of onset of TEAE – study drug start date + 1) /365.25

If, for a subject, the selected treatment emergent adverse event didn't occur then the time at risk, for the analysis phases according to randomized treatment, will be censored at the minimum of either date of death, last contact date per EoS page, or randomized drug stop date + 140 days. For each selected treatment emergent AE, the exposure adjusted incidence rate will be calculated as:

Incidence rate [1/100 Subject years (pt-yrs)] = 100 \* number of subjects with AE /Total AE-specific time at risk [subject years].

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the exposure adjusted incidence rates (per 100 subject years) as well as the number of patients with AEs, and not on the number of AEs. System organ classes (if applicable) will be sorted according to the standard sort order specified by the EMA. Preferred terms (if applicable) will be sorted by total frequency (within system organ class) across all treatment arms, or, if a total column across all arms is not foreseen in the table, by total frequency (within system organ class) within the BI arm.

For details on summarization of AE data, please refer to "Handling and summarization of adverse event data for clinical trial reports and integrated summaries" (7) [001-MCG-156] and *BI-KMED-BDS-HTG-0035*: "Handling of missing and incomplete AE dates" (4).

The analysis of AEs will be based on the concept of treatment emergent AEs. Since only the start date of an AE is collected (without start time), any AE occurrence on the same day as the first BI 655130 administration will be assigned to the on-treatment period.

An overall summary of AEs will be presented by treatment. This overall summary will include summary statistics for the class of other significant AEs according to sponsor definition based on ICH E3 and for the class of AESIs.

The following are considered as AESIs (see CTP section 5.3.6.1):

- Infusion reactions including anaphylactic reaction
- Cytokine release syndrome
- Severe bacterial, fungal, and viral infections
- Infection with or reactivation of mycobacterium tuberculosis,
- Opportunistic infections
- Lymphoproliferative disorders
- Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o an elevation of AST and/or ALT  $\geq$ 3 fold ULN combined with an elevation of total bilirubin  $\geq$ 2 fold ULN measured in the same blood draw sample, and/or
- o marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN.

The investigator identified AESI will be captured from the eCRF and reported in the "Investigator reported AESI" table. In addition, User-defined Adverse Event Concepts (UDAEC) identified through specific search criteria will be reported separately (see <u>Table 7.8.1: 1</u>). For these displays, separate tables will be created for each AESI category wherein frequencies by treatment group will be given.

Trial No: 1368-0010 - 3.0 (Final)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.8.1: 1 Project MEDDRA search criteria for User Defined Adverse Events Concepts

| User Defined Adverse<br>Event Concepts | Categories |
|---|---|
| Infusion/Systemic | Narrow SMQ "Anaphylactic reaction" |
| hypersensitivity reactions | Narrow SMQ "Angioedema" |
| including anaphylactic reactions | Narrow SMQ "Hypersensitivity" |
| Severe infections (according to RCTC grading) | SOC Infections and infestations of at least severe RCTC grade, by HLGT |
| Opportunistic and | BIcMQ "Infections": |
| mycobacterium tuberculosis infections | Narrow sub-search 8 "Opportunistic infections including Tuberculosis related terms" |
| Tuberculosis related terms | BIcMQ "Infections": |
| | Narrow sub-search 8.2 "Tuberculosis related terms" |
| | HLT "Tuberculosis infections" |
| Malignant tumours | (SMQ "Malignancies" – not for display) |
| | (Sub-SMQ "Malignant or unspecified tumours" – not for display) |
| | Narrow Sub-SMQ "Malignant tumours" |
| | Sub-SMQ "Haematological malignant tumours" |
| | Sub-SMQ "Non-Haematological malignant |
| | tumours" |

Based on the specification provided in ICH E3 (9), the sponsor has defined AEs which are to be classified as 'other significant'. For the current trial, these will include those non-serious AEs which were reported with 'action taken = Drug Withdrawn' or 'action taken = Dose Reduced',

The exposure-adjusted incidence rate and frequency of patients with AEs will be summarised by treatment, primary system organ class, and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for patients with SAEs, patients with AESIs, patients with AE leading to discontinuation of the trial, patients with other significant AEs and User-defined Adverse Event Concepts (UDAEC) (see <u>Table 7.8.1: 1</u>). AEs will also be summarized by maximum intensity based on the RCTC measure (see <u>Section 5.4.1</u>).

For disclosure of AE data on ClinicalTrials.gov, the frequency of patients with non-serious AEs occurring with an incidence of greater than 5% (in preferred terms) will be summarised by treatment, primary system organ class and preferred term. The frequency of patients with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of non-serious AEs with an incidence of greater than 5% (in preferred terms) and the frequency of SAEs will be summarised.

# 7.8.2 **Laboratory data**

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (8). Note that data from the central laboratory will be used for all displays described below, unless otherwise specified.

For continuous safety laboratory parameters, normalized values will be derived. Normalisation means transformation to a standard unit and to a standard reference range. The process of normalisation, handling of repeat values at the same visit for by-visit displays, as well as standard analyses for safety laboratory data are all described in the BI guidance for the Display and Analysis of Laboratory Data (8). All analyses considering multiple times of the ULN (as described below) will be based on standardized and not normalized values. For continuous safety laboratory parameters, differences to baseline will be calculated.

Only patients with at least one available post-baseline value will be included in the analysis of an individual laboratory parameter. All individual laboratory data will be listed. Values outside the reference range will be flagged.

Descriptive statistics of laboratory values over time (using on treatment data) and for the difference from baseline (see Section 6.7) will be based upon standardized values and provided by visit, including summaries of the last value on treatment, the minimum value on treatment, and the maximum value on treatment. Graphical displays via box plots will be produced for the change from baseline over time for each continuous laboratory endpoint.

Laboratory values will be compared to their reference ranges. Shift tables will be provided for the number of patients with a specific RCTC grade at baseline versus the grade at the last measurement on treatment, as well as the worst grade on treatment. These analyses will be based on standardized laboratory values.

Potentially clinically significant on-treatment abnormalities will be identified based on BI standard rules, which are based on normalized converted lab values, i.e., using the International System of Units. These rules will be listed in the SDL appendix of the CTR. Frequency tables will summarize the number of patients with potentially clinically significant abnormalities for patients without a possibly clinically significant abnormality at baseline. A separate listing will present potentially clinically significant abnormal lab values. If there exists at least one lab value with a clinically significant abnormality within a functional lab group, then for each functional lab group all patient's lab values will be listed.

The frequency of patients with AST or ALT elevations  $\geq 3x$  ULN,  $\geq 5x$  ULN,  $\geq 10x$  ULN, and  $\geq 20x$  ULN will be displayed based on standardized laboratory values. To support analyses of liver related adverse drug effects, the frequency of patients with AST and/or ALT  $\geq 3x$  ULN combined with a total bilirubin  $\geq 2x$  ULN in a 30-day period after AST/ALT elevation will be displayed, stratified by alkaline phosphatase  $\leq 2x$  ULN and  $\geq 2x$  ULN (a

patient can potentially be in both alkaline phosphatase strata in case of multiple AST/ALT and bilirubin elevations). The start of the 30-day time span is triggered by each liver enzyme elevation above the defined thresholds. This analysis will be based on on-treatment standardized laboratory values.

A graphical analysis of the ALT and total bilirubin during the on-treatment period will also be performed; the so called eDISH plot. In the graph, for each subject, the peak total bilirubin is presented as a fold increase over the ULN against the peak ALT as a fold increase over the ULN, on a log10 scale. The measurements displayed or total bilirubin and ALT may, or may not, occur on the same date. Two reference lines, 2x ULN for total bilirubin and 3x ULN for ALT, are drawn onto the graph in order to divide the plane into four quadrants. Normal cases are in the lower left quadrant, potential DILI cases are in the upper right quadrant (Hy's Law quadrant), while the lower right quadrant is known as the Temple's corollary range (ALT  $\geq$  3x ULN and total bilirubin < 2x ULN).

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

# 7.8.3 Vital signs

The analyses of vital signs (blood pressure, pulse rate, body temperature, and body weight) will be descriptive in nature.

Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided by treatment. At each on-treatment time-point, three assessments will be presented: the pre-dose measurement, the +5 minutes post-dose measurement, and the +2 hours post-dose measurement; change from baseline refers to the original baseline value. The summary will include additionally, the last value, the minimum value, and the maximum value during the on-treatment period presented for each of the three visit measurement times separately (see Table 6.1: 1 for the definition of the on-treatment period). Graphical displays via box plots will be produced for the change from baseline over time for each continuous vital sign endpoint.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### 7.8.4 **ECG**

Abnormal findings in 12-lead ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

No separate listing or analysis of ECG data will be prepared.

# 7.8.5 **Others**

The frequency and percentage of patients with ADA to BI 655130 will be presented by visit. ADA will be analysed descriptively. A potential effect of ADA on PK and safety may be evaluated.

# 8. REFERENCES

- 1 *CPMP/ICH/363/96*: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9; Note For Guidance on Statistical Principles for Clinical Trials, current version
- 2 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON
- 3 *BI-KMED-COPS-TMP-0001:* "Important Protocol Deviation (iPD) log", current version; IDEA for CON
- 4 *BI-KMED-BDS-HTG-0035*: "Handling of missing and incomplete AE dates", current version; IDEA for CON
- 5 001-MCS-36-472\_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON
- 6 001-MCS-36-472\_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON
- 7 001-MCG-156: "Handling and summarisation of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON
- 8 *BI-KMED-BDS-HTG-0042*: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON
- 9 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version
- 10 *BI-KMED-BDS-HTG-0045:* "Standards for Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON
- 11 001-MCS-36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON
- 12 Devlin N, Shah K, Feng Y, Mulhern B, van Hout B. Valuing Health-Related Quality of Life: An EQ-5D-5L Value Set for England. OHE Research Paper 16/01. London: Office of Health Economics; 2016 [R17-3268]
- SAS/STAT(R) 9.2 User's Guide, Second Edition. http://support.sas.com/documentation/cdl/en/statug/63033/HTML/default/viewer.ht m#statug lifetest a0000000260.htm (retrieved 16-May-2018)
- 14 Brown LD, Cai TT, DasGupta A. Confidence intervals for a binomial proportion and asymptotic expansions. Ann Statistics 30, 160-201, 2002 [R12-3710]

# **Boehringer Ingelheim**

**Trial No: 1368-0010 – 3.0 (Final)** 


Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Newcombe R.G. Interval estimation for the difference between independent proportions: Comparison of eleven methods. Stat Methods Med Res 17, 873-890 1998 [R08-4386]
- Marchal-Bressenot A, Salleron J, Boulagnon-Rombi C, et al.: Development and validation of the Nancy histological index for UC . Gut 2017; 66:43–49. [R18-1193]



















#### **10. HISTORY TABLE**

History table Table 10: 1

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial 1.0 | 19-May-2017 | | None | First approved version before first patient in. |
| 1.1 (Stable TSAP) | 01-Aug-2017 | | (multiple) | Stable TSAP after team comments at TSAP walkthrough, basis for initial programming. Various additions, including: Code for Reeve's method added; text for IBDQ and EQ-5D was amended. Analyses of biomarkers was removed to be shifted to a separate BM-SAP. |
| 2.0 | 26-Aug-2019 | | (all) | This is the final version of core TSAP |
| 3.0 | 04-Mar-2020 | | (all) | This is the revised TSAP due to early termination of the study. |